CLINICAL TRIAL: NCT00413608
Title: Influence of CYP2C19 Genetic Variants on Clopidogrel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department Clinical Research of developpement
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060309
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
Keywords: Human; Adults; Male; Alleles; Genotype; Platelet Aggregation/drug effects; Platelet Aggregation Inhibitors/*pharmacology; Platelet Function Tests; Pharmacogenetics; *Polymorphism, Genetic; Ticlopidine/*analogs & derivatives/pharmacology; Healthy subjects
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Clopidogrel
  Interventions: Drug: Clopidogrel
- 2 (Experimental): Clopidogrel
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel

SUMMARY:
To test pharmacodynamic response to clopidogrel 150mg once daily during 7 days in healthy subjects carriers of a mutated allele (*2) associated with CYP2C19 deficiency and non responders to the usual regimen of 75 mg once daily

DETAILED DESCRIPTION:
Thirty individuals genotyped for specific variants of 2C19 cytochrome and P2Y12 platelet ADP receptor will receive during one week a daily dose of 75 mg of clopidogrel. Depending on their pharmacodynamic response to this dose of clopidogrel, subjects will be affiliated to two groups, "good responders" and "bad responders". After a wash-out period, "bad responders" will receive a double dose of clopidogrel, while the "good responders" will receive 75 mg of clopidogrel, associated with a CYP2C19 inhibitor. Such study will allow to evaluate both the impact of raising daily dose of clopidogrel in patients with defected variants of 2C19 and potential interactions of clopidogrel with other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged 18 to 35, non smoker, of caucasian origin
* Compatible 2C19 and P2Y12 genotypes
* Weight 60 kg to 100 kg, and normal BMI
* Standard laboratory investigations normal
* Negative testing for HIV infection and B and C hepatitis
* Basal platelet agregation testing normal
* EKG, blood pressure and cardiac frequency in normal range
* Ability to understand, follow and sign the protocol

Exclusion Criteria:

* Evolutive medical affection, even treated
* Medical history of allergic response to medication or other, peptic ulcer, or known hemorrhagic disorder
* Laboratory testing out of normal range
* Subjects practicing violent sports
* Unability to understand or follow the protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Inhibition platelet activity index (ADP induced aggregation) measured between | during 7 days

SECONDARY OUTCOMES:
Clopidogrel and metabolites pharmacokinetics and relation to dynamics | during 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Sébastien HULOT, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Result] Hulot JS, Bura A, Villard E, Azizi M, Remones V, Goyenvalle C, Aiach M, Lechat P, Gaussem P. Cytochrome P450 2C19 loss-of-function polymorphism is a major determinant of clopidogrel responsiveness in healthy subjects. Blood. 2006 Oct 1;108(7):2244-7. doi: 10.1182/blood-2006-04-013052. Epub 2006 Jun 13. PMID 16772608